CLINICAL TRIAL: NCT00086190
Title: Study of Antidepressants in Parkinson's Disease
Acronym: SAD-PD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Irene Richard, Irene Richard, MD, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01NS046487 (NIH)
Record Dates: First submitted 2004-06-28; First posted 2004-06-29 (Estimated); Results first posted 2013-01-04 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Parkinson Disease; Depression
Keywords: Parkinson disease; depression; Parkinson's disease; paroxetine; venlafaxine; antidepressant
MeSH Terms: conditions — Parkinson Disease; Depression | interventions — Paroxetine; Venlafaxine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- paroxetine (Active Comparator): Paroxetine and venlafaxine will be compared to placebo over 12 weeks.
  Interventions: Drug: paroxetine
- venlafaxine extended release (Active Comparator): Paroxetine and venlafaxine will be compared to placebo over 12 weeks.
  Interventions: Drug: venlafaxine
- placebo (Placebo Comparator): Paroxetine and venlafaxine will be compared to placebo over 12 weeks.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: paroxetine — Paroxetine 10 mg tablets or matching placebo given once a day for the first two weeks. If depression is not being effectively treated then the paroxetine or matching placebo will be increased to 20 mg, followed by a 10 mg increase every two weeks (if tolerated). Dosage for this study will not exceed 40 mg.
  Other Names: Paxil
  Arms: paroxetine
Drug: venlafaxine — Venlafaxine XR 37.5 mg capsules or matching placebo given once a day for the first two weeks. If depression is not being effectively treated then the venlafaxine XR capsules or matching placebo will be increased to 75 mg followed by 75 mg increments every 2 weeks (if tolerated). Dosage for this study will not exceed 225 mg.
  Other Names: Effexor XR
  Arms: venlafaxine extended release
Other: placebo — an inactive substance
  Arms: placebo

SUMMARY:
The purpose of this study is to find out if two antidepressant medications, paroxetine and venlafaxine, can help control depression in Parkinson's disease, and if these medications affect the motor symptoms of Parkinson's disease such as tremor, stiffness, slowness, and balance.

DETAILED DESCRIPTION:
Nearly 50 percent of individuals with Parkinson's disease (PD) suffer from depression-a condition that causes disability and can reduce quality of life. The University of Rochester Medical Center is conducting a research study of antidepressant medications to find out more about how to treat depression in PD. Antidepressant medications have not been adequately studied in persons with PD.

The purpose of this study is to find out if the antidepressant medications paroxetine and venlafaxine can help control depression in PD and whether or not these medications affect the motor symptoms of PD such as tremor, stiffness, slowness, and balance.

This is a randomized, double blind, placebo-controlled, 12-week study of paroxetine immediate release (Paxil) and venlafaxine extended release (Effexor XR). Paroxetine and venlafaxine XR are drugs that have been approved by the Food and Drug Administration (FDA) and are available by prescription. Paroxetine and venlafaxine XR have been shown to be effective in treating depression in the general population. Two hundred, twenty-eight persons will be enrolled among 15 medical centers throughout the United States and Canada. Each person will participate in the trial for 12 weeks. Each participant will be randomly assigned to take either paroxetine or venlafaxine, or a placebo.

ELIGIBILITY:
Inclusion Criteria:

To be eligible you must be:

* 30 years old or older
* diagnosed with Parkinson's disease
* experiencing symptoms of depression such as sadness, decreased energy, or problems sleeping

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2005-06; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irene Richard, MD, Principal Investigator — University of Rochester; William McDonald, MD, Principal Investigator — Co-Principal Investigator--Emory University School of Medicine
Locations (18):
- United States (15):
  - University of California San Francisco, San Francisco, California
  - University of Florida, Gainesville, Florida
  - University of Miami, Miami, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - University of Kentucky, Lexington, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - University of Maryland, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Dept. of Neurology E/KS 430, 330 Brookline Avenue, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - University of Rochester, Rochester, New York
  - Medical University of Ohio, Toledo, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - University of Tennessee-Memphis, Memphis, Tennessee
  - Baylor College of Medicine, 6550 Fannin, Suite 1801, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
- Canada (2):
  - London Health Sciences Centre, University Campus Room A10-325, 339 Windermere Road, London, Ontario
  - Hotel-Dieu Hospital-CHUM, Montreal, Quebec
- University of Puerto Rico, San Juan, Puerto Rico

REFERENCES:
- [Background] Dooneief G, Mirabello E, Bell K, Marder K, Stern Y, Mayeux R. An estimate of the incidence of depression in idiopathic Parkinson's disease. Arch Neurol. 1992 Mar;49(3):305-7. doi: 10.1001/archneur.1992.00530270125028. PMID 1536634
- [Background] Liu CY, Wang SJ, Fuh JL, Lin CH, Yang YY, Liu HC. The correlation of depression with functional activity in Parkinson's disease. J Neurol. 1997 Aug;244(8):493-8. doi: 10.1007/s004150050131. PMID 9309555
- [Background] Kuopio AM, Marttila RJ, Helenius H, Toivonen M, Rinne UK. The quality of life in Parkinson's disease. Mov Disord. 2000 Mar;15(2):216-23. doi: 10.1002/1531-8257(200003)15:23.0.co;2-#. PMID 10752569
- [Background] Phillips P. Keeping depression at bay helps patients with Parkinson disease. JAMA. 1999 Sep 22-29;282(12):1118-9. No abstract available. PMID 10501101
- [Background] Global Parkinson's Disease Survey (GPDS) Steering Committee.. Factors impacting on quality of life in Parkinson's disease: results from an international survey. Mov Disord. 2002 Jan;17(1):60-7. doi: 10.1002/mds.10010. PMID 11835440
- [Background] Menza M, Dobkin RD, Marin H, Mark MH, Gara M, Buyske S, Bienfait K, Dicke A. A controlled trial of antidepressants in patients with Parkinson disease and depression. Neurology. 2009 Mar 10;72(10):886-92. doi: 10.1212/01.wnl.0000336340.89821.b3. Epub 2008 Dec 17. PMID 19092112
- [Background] Devos D, Dujardin K, Poirot I, Moreau C, Cottencin O, Thomas P, Destee A, Bordet R, Defebvre L. Comparison of desipramine and citalopram treatments for depression in Parkinson's disease: a double-blind, randomized, placebo-controlled study. Mov Disord. 2008 Apr 30;23(6):850-7. doi: 10.1002/mds.21966. PMID 18311826
- [Background] Yeragani VK, Roose S, Mallavarapu M, Radhakrishna RK, Pesce V. Major depression with ischemic heart disease: effects of paroxetine and nortriptyline on measures of nonlinearity and chaos of heart rate. Neuropsychobiology. 2002;46(3):125-35. doi: 10.1159/000066390. PMID 12422059
- [Background] Yeragani VK, Pesce V, Jayaraman A, Roose S. Major depression with ischemic heart disease: effects of paroxetine and nortriptyline on long-term heart rate variability measures. Biol Psychiatry. 2002 Sep 1;52(5):418-29. doi: 10.1016/s0006-3223(02)01394-x. PMID 12242058
- [Background] Nelson JC, Kennedy JS, Pollock BG, Laghrissi-Thode F, Narayan M, Nobler MS, Robin DW, Gergel I, McCafferty J, Roose S. Treatment of major depression with nortriptyline and paroxetine in patients with ischemic heart disease. Am J Psychiatry. 1999 Jul;156(7):1024-8. doi: 10.1176/ajp.156.7.1024. PMID 10401446
- [Background] Simons JA. Fluoxetine in Parkinson's disease. Mov Disord. 1996 Sep;11(5):581-2. doi: 10.1002/mds.870110517. No abstract available. PMID 8866503
- [Background] Steur EN. Increase of Parkinson disability after fluoxetine medication. Neurology. 1993 Jan;43(1):211-3. doi: 10.1212/wnl.43.1_part_1.211. PMID 8423889
- [Background] Jimenez-Jimenez FJ, Tejeiro J, Martinez-Junquera G, Cabrera-Valdivia F, Alarcon J, Garcia-Albea E. Parkinsonism exacerbated by paroxetine. Neurology. 1994 Dec;44(12):2406. doi: 10.1212/wnl.44.12.2406. No abstract available. PMID 7991139
- [Background] Salzman C. Pharmacologic treatment of depression in the elderly. J Clin Psychiatry. 1993 Feb;54 Suppl:23-8. PMID 8444831
- [Background] Altamura AC, De Novellis F, Guercetti G, Invernizzi G, Percudani M, Montgomery SA. Fluoxetine compared with amitriptyline in elderly depression: a controlled clinical trial. Int J Clin Pharmacol Res. 1989;9(6):391-6. PMID 2699465
- [Background] Feighner JP, Boyer WF, Meredith CH, Hendrickson G. An overview of fluoxetine in geriatric depression. Br J Psychiatry Suppl. 1988 Sep;(3):105-8. No abstract available. PMID 3074861
- [Background] Cohn CK, Shrivastava R, Mendels J, Cohn JB, Fabre LF, Claghorn JL, Dessain EC, Itil TM, Lautin A. Double-blind, multicenter comparison of sertraline and amitriptyline in elderly depressed patients. J Clin Psychiatry. 1990 Dec;51 Suppl B:28-33. PMID 2258379
- [Background] Dubovsky S. Geriatric Neuropsychopharmacology. In: Coffey C, Cummings J, eds. Textbook of Geriatric Neuropsychiatry. Washington, DC: American Psychiatric Press, 1994:595-631.
- [Background] Dunner DL, Cohn JB, Walshe T 3rd, Cohn CK, Feighner JP, Fieve RR, Halikas JP, Hartford JT, Hearst ED, Settle EC Jr, et al. Two combined, multicenter double-blind studies of paroxetine and doxepin in geriatric patients with major depression. J Clin Psychiatry. 1992 Feb;53 Suppl:57-60. PMID 1531827
- [Background] Guillibert E, Pelicier Y, Archambault JC, Chabannes JP, Clerc G, Desvilles M, Guibert M, Pagot R, Poisat JL, Thobie Y. A double-blind, multicentre study of paroxetine versus clomipramine in depressed elderly patients. Acta Psychiatr Scand Suppl. 1989;350:132-4. doi: 10.1111/j.1600-0447.1989.tb07192.x. No abstract available. PMID 2530766
- [Background] Hirschfeld RM. Efficacy of SSRIs and newer antidepressants in severe depression: comparison with TCAs. J Clin Psychiatry. 1999 May;60(5):326-35. doi: 10.4088/jcp.v60n0511. PMID 10362442
- [Background] Entsuah AR, Huang H, Thase ME. Response and remission rates in different subpopulations with major depressive disorder administered venlafaxine, selective serotonin reuptake inhibitors, or placebo. J Clin Psychiatry. 2001 Nov;62(11):869-77. doi: 10.4088/jcp.v62n1106. PMID 11775046
- [Background] Gentil V, Kerr-Correa F, Moreno R, D'Arrigo Busnello E, De Campos JA, Juruena MF, Lafer B, Moreno DH, De Cassia Rodrigues RL, Tiosso A, Benedictis E. Double-blind comparison of venlafaxine and amitriptyline in outpatients with major depression with or without melancholia. J Psychopharmacol. 2000 Mar;14(1):61-6. doi: 10.1177/026988110001400108. PMID 10757255
- [Background] Applebaum PS, Grisso T. MacCAT-CR: MacArthur Competence Assessment Tool for Clinical Research. Sarasota, FL: Professional Resource Press, 2001.
- [Background] American Psychiatric Association. Diagnostic and Statistical Manual of Mental Disorders, 4th ed. Washington, DC, 1994.
- [Background] Spitzer RL, Gibbon M, Williams JBW. Structured clinical interview for Axis I DSM-IV disorders: Biometrics Research Department. New York State Psychiatric Institute 1994.
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] HAMILTON M. A rating scale for depression. J Neurol Neurosurg Psychiatry. 1960 Feb;23(1):56-62. doi: 10.1136/jnnp.23.1.56. No abstract available. PMID 14399272
- [Background] Montgomery SA, Asberg M. A new depression scale designed to be sensitive to change. Br J Psychiatry. 1979 Apr;134:382-9. doi: 10.1192/bjp.134.4.382. PMID 444788
- [Background] Beck AT, Steer RA, Ball R, Ranieri W. Comparison of Beck Depression Inventories -IA and -II in psychiatric outpatients. J Pers Assess. 1996 Dec;67(3):588-97. doi: 10.1207/s15327752jpa6703_13. PMID 8991972
- [Background] Yesavage JA, Brink TL, Rose TL, Lum O, Huang V, Adey M, Leirer VO. Development and validation of a geriatric depression screening scale: a preliminary report. J Psychiatr Res. 1982-1983;17(1):37-49. doi: 10.1016/0022-3956(82)90033-4. PMID 7183759
- [Background] Conners CK, Barkley RA. Rating scales and checklists for child psychopharmacology. Psychopharmacol Bull. 1985;21(4):809-43. No abstract available. PMID 4089107
- [Background] Fahn S, Elton RL. Unified Parkinson's Disease Rating Scale. In: Fahn S, Marsden CD, Calne DB, Goldstein M, eds. Recent Developments in Parkinson's Disease. Florham Park, NJ: MacMillan Healthcare Information, 1992:153-163.
- [Background] Uc EY, McDermott MP, Marder KS, Anderson SW, Litvan I, Como PG, Auinger P, Chou KL, Growdon JC; Parkinson Study Group DATATOP Investigators. Incidence of and risk factors for cognitive impairment in an early Parkinson disease clinical trial cohort. Neurology. 2009 Nov 3;73(18):1469-77. doi: 10.1212/WNL.0b013e3181bf992f. PMID 19884574
- [Background] Lachin JM. Introduction to sample size determination and power analysis for clinical trials. Control Clin Trials. 1981 Jun;2(2):93-113. doi: 10.1016/0197-2456(81)90001-5. PMID 7273794
- [Background] Little RJA, Rubin DB. Statistical Analysis with Missing Data, Second Edition. Hoboken: John Wiley and Sons, 2002.
- [Background] McDonald WM, Holtzheimer PE, Haber M, Vitek JL, McWhorter K, Delong M. Validity of the 30-item geriatric depression scale in patients with Parkinson's disease. Mov Disord. 2006 Oct;21(10):1618-22. doi: 10.1002/mds.21023. PMID 16817205
- [Background] Okun MS, Fernandez HH. Will tricyclic antidepressants make a comeback for depressed Parkinson disease patients? Neurology. 2009 Mar 10;72(10):868-9. doi: 10.1212/01.wnl.0000338145.24512.02. Epub 2008 Dec 17. No abstract available. PMID 19092111
- [Background] Brunoni AR, Lopes M, Kaptchuk TJ, Fregni F. Placebo response of non-pharmacological and pharmacological trials in major depression: a systematic review and meta-analysis. PLoS One. 2009;4(3):e4824. doi: 10.1371/journal.pone.0004824. Epub 2009 Mar 18. PMID 19293925
- [Background] Senn S, Julious S. Measurement in clinical trials: a neglected issue for statisticians? Stat Med. 2009 Nov 20;28(26):3189-209. doi: 10.1002/sim.3603. PMID 19455540

RESULTS

PARTICIPANT FLOW:
Recruitment Details: SAD-PD enrolled 115 participants from 20 centers in the US, Canada, and Puerto Rico from June 2005 through March 2009. Participants were recruited from movement disorder clinics. Eligible participants included men and women 30 years and older who were diagnosed with idiopathic PD, without dementia and who met depression criteria.
Groups:
- Paroxetine: Optimal paroxetine dosage was determined on a per patient basis. The mean dosage at week 12 was 24 +/- 11 mg/day.
- Venlafaxine Extended Release: Optimal venlafaxine extended release dosage was determined on a per patient basis. The mean dosage at week 12 was 121 +/- 75 mg/day.
- Placebo: Placebo was made to match treatment options.
Period: Overall Study
Arm/Group | Paroxetine | Venlafaxine Extended Release | Placebo
Started | 42 | 34 | 39
Completed | 34 | 30 | 33
Not Completed | 8 | 4 | 6
Not completed — Adverse Event | 6 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 2 | 2
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Moved | 1 | 0 | 0
Not completed — Worsening depression | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paroxetine | Venlafaxine Extended Release | Placebo | Total
Number analyzed (Participants) | 42 | 34 | 39 | 115
Age Continuous [Mean (Standard Deviation); unit: years] | 65.2 (9.8) | 62.5 (11.4) | 62.7 (11.0) | 63.5 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 15 | 16 | 42
  Male | 31 | 19 | 23 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 4 | 12
  Not Hispanic or Latino | 38 | 30 | 35 | 103
  Unknown or Not Reported | 0 | 0 | 0 | 0
Education beyond High School [Number; unit: participants]
  Beyond High School | 35 | 27 | 27 | 89
  Not beyond High School | 7 | 7 | 12 | 26
Marriage [Number; unit: participants]
  Married | 27 | 27 | 28 | 82
  Not married | 15 | 7 | 11 | 33
Major Depression [Number; unit: participants]
  Yes | 29 | 22 | 22 | 73
  No | 13 | 12 | 17 | 42
Past Antidepressant Use [Number; unit: participants]
  Yes | 3 | 2 | 5 | 10
  No | 39 | 32 | 34 | 105
HAM-D Score [Mean (Standard Deviation); unit: Hamilton Depression Score] — Hamilton Depression Rating Scale. Ranges from 0-50. Higher scores represent more significant depression. Mild depression ranges from 8-13, moderate depression from 14-18, severe 19-22 and very severe any score over 23.
  Hamilton Depression Score | 22.2 (6.5) | 21.2 (6.0) | 21.4 (4.8) | 21.6 (5.8)
MADRS Score [Mean (Standard Deviation); unit: Score] — Montgomery-Asberg Depression Rating Scale. Range 0-60. Higher score indicates more severe depression. 0-6 normal, 7-19 mild depression, 20-34 moderate depression, greater than 34 severe depression.
  Score | 21.0 (6.8) | 19.4 (7.9) | 19.9 (5.9) | 20.1 (6.9)
GDS Score [Mean (Standard Deviation); unit: Score] — Geriatric Depression Scale. Range 0-30. Higher score indicates more severe depression. 0-9 normal, 10-19 mild depression, 20-30 severe depression.
  Score | 15.5 (6.2) | 15.1 (5.8) | 15.0 (4.9) | 15.2 (5.6)
BDI-II Score [Mean (Standard Deviation); unit: Score] — Beck Depression Inventory II. Range 0-63. Higher score indicates more severe depression. 0-13 minimal depression, 14-19 mild depression, 20-28 moderate depression, 29-63 severe depression.
  Score | 17.2 (9.2) | 17.1 (9.1) | 17.5 (7.4) | 17.3 (8.6)
Years since PD Onset [Mean (Standard Deviation); unit: Years] | 6.7 (5.8) | 7.4 (4.2) | 7.0 (3.8) | 7.0 (4.6)
Years since PD Diagnosis [Mean (Standard Deviation); unit: Years] | 5.2 (5.9) | 4.7 (3.7) | 4.9 (3.6) | 4.9 (4.4)
Hoehn and Yahr Stage [Number; unit: Participants] — As the stage rating increases, the severity of the disease increases. Ranges from 1.0 to 5.0.
  Participants
    1.0-1.5 (Unilateral Parkinson's Disease) | 3 | 0 | 3 | 6
    2.0-2.5 (Mild Bilateral Parkinson's Disease) | 32 | 29 | 31 | 92
    3.0-4.0 (Moderate to Severe Bilateral Parkinson's) | 7 | 5 | 5 | 17
UPDRS Score [Mean (Standard Deviation); unit: Score] — Unified Parkinson's Disease Rating Scale. Higher score indicates more severe Parkinson's disease symptoms. Total maximum = 176. Mental maximum = 52, Activities of Daily Living maximum = 52, Motor maximum = 72. Minimum score = 0.
  Score
    Mental | 4.8 (2.4) | 5.2 (1.9) | 4.6 (2.0) | 4.9 (2.1)
    Activities of Daily Living | 27.3 (9.6) | 26.8 (12.3) | 26.4 (11.5) | 26.8 (11.1)
    Motor | 10.6 (6.7) | 11.4 (7.4) | 10.8 (5.5) | 10.9 (6.5)
    Total | 42.7 (14.9) | 43.1 (19.0) | 41.7 (15.9) | 42.5 (16.6)
Schwab/England Activities of Daily Living Score ("On") [Mean (Standard Deviation); unit: Score] — Schwab and England Activities of Daily Living Scale (S/E ADL). Range 0-100%. Higher percentage indicates higher level of function and lower impact of disease on life activities.
  Score | 82.9 (11.2) | 80.3 (14.6) | 80.8 (13.4) | 81.3 (13.1)
Motor Fluctuations [Number; unit: Participants]
  Yes | 25 | 20 | 24 | 69
  No | 17 | 14 | 15 | 46
PDQ-39 Total [Mean (Standard Deviation); unit: Score on PDQ-39 Questionnaire] — Parkinson's Disease Questionnaire (PDQ-39) Total. Range 0-100. Lower score indicates a better perceived health status.
  Score on PDQ-39 Questionnaire | 36.8 (16.3) | 37.2 (15.6) | 39.6 (14.8) | 37.9 (15.6)
Short Form-36 Health Survey Scores [Mean (Standard Deviation); unit: Score] — Short Form 36 Health Survey. Range 0-100. Higher score indicates a better perceived quality of life.
  Score
    Physical Component Summary | 37.5 (9.3) | 36.2 (10.3) | 37.1 (10.4) | 36.9 (10)
    Mental Component Summary | 41.4 (8.8) | 38.3 (10.1) | 40.0 (9.3) | 39.9 (9.4)
Snaith CAS [Mean (Standard Deviation); unit: Score] — Snaith Clinical Anxiety Scale. Range 0-21. Higher scores indicate increased anxiety. Score greater than 8 indicates clinical anxiety.
  Score | 6.7 (3.9) | 7.8 (4.5) | 7.5 (4.3) | 7.3 (4.2)
Mini Mental State Examination Score [Mean (Standard Deviation); unit: Score] — Mini Mental State Examination (MMSE). Range 0-30. Higher score indicates better cognitive status. Score less than 9 = severe cognitive impairment, 10-20 moderate impairment, 21-24 mild impairment, 25 and greater considered normal.
  Score | 28.7 (1.4) | 28.9 (1.8) | 28.5 (1.5) | 28.7 (1.6)
BPRS Score [Mean (Standard Deviation); unit: Score] — Brief Psychiatric Rating Scale. Maximum score 126, minimum score 0. Higher score indicates greater psychiatric difficulties.
  Score | 33.6 (10.7) | 35.7 (8.9) | 34.4 (9.3) | 34.6 (9.6)
Treatment of PD - Levodopa [Number; unit: Participants] — Participants taking Levodopa for treatment of Parkinson's Disease.
  Participants
    Treatment - Yes | 38 | 27 | 32 | 97
    Treatment - No | 4 | 7 | 7 | 18
Treatment of PD - Agonist [Number; unit: Participants] — Participants taking Agonist for treatment of Parkinson's Disease.
  Participants
    Treatment - Yes | 17 | 13 | 12 | 42
    Treatment - No | 25 | 21 | 27 | 73
Treatment for PD - Catechol O-methyltransferase Inhibitor [Number; unit: Participants] — Participants taking Catechol O-methyltransferase (COMT) Inhibitor for treatment of Parkinson's Disease.
  Participants
    Treatment - Yes | 9 | 9 | 11 | 29
    Treatment - No | 33 | 25 | 28 | 86
Treatment of PD - Amantadine [Number; unit: Participants] — Participants taking Amantadine for treatment of Parkinson's Disease.
  Participants
    Treatment - Yes | 6 | 4 | 6 | 16
    Treatment - No | 36 | 30 | 33 | 99
Treatment of PD - Anticholinergic [Number; unit: Participants] — Participants taking Anticholinergic for treatment of Parkinson's Disease.
  Participants
    Treatment - Yes | 3 | 4 | 3 | 10
    Treatment - No | 39 | 30 | 36 | 105

OUTCOME MEASURES:

1. Primary Outcome: Change in Hamilton Depression Rating Scale (HAM-D) Scores
Description: Change in Hamilton Rating Scale for Depression over 12 weeks. Hamilton Depression Rating Scale ranges from 0-50. Higher scores represent more significant depression. Mild depression ranges from 8-13, moderate depression from 14-18, severe 19-22 and very severe any score over 23.
Time Frame: from the beginning (0 weeks) to end (12 weeks) of the double-blind phase
Population: 115 subjects were randomized to receive either Paroxetine, Venlafaxine ER or placebo. All randomized participants were included in analysis, in accordance to intention-to-treat principle.
Measure: Mean (Standard Deviation); unit: Change in HAM-D score
Groups:
- Paroxetine: Mean change in outcome measure from baseline for participants taking paroxetine.
- Venlafaxine Extended Release: Mean change in outcome measure from baseline for participants taking venlafaxine ER.
- Placebo: Mean change in outcome measure from baseline for participants taking placebo.
Arm/Group | Paroxetine | Venlafaxine Extended Release | Placebo
Number analyzed (Participants) | 42 | 34 | 39
Change in HAM-D score | -13.0 (1.3) | -11.0 (1.4) | -6.8 (1.3)

2. Secondary Outcome: Change in Montgomery-Asberg Depression Rating Scale (MADRS)
Description: Montgomery-Asberg Depression Rating Scale ranges from 0-60. Higher score indicates more severe depression. 0-6 normal, 7-19 mild depression, 20-34 moderate depression, greater than 34 severe depression.
Time Frame: from the beginning (0 weeks) to end (12 weeks) of the double-blind phase
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Change in MADRS score
Arm/Group | Paroxetine | Venlafaxine Extended Release | Placebo
Number analyzed (Participants) | 42 | 34 | 39
Change in MADRS score | -13.6 (1.2) | -10.9 (1.3) | -6.6 (1.2)

3. Secondary Outcome: Change in Beck Depression Inventory II (BDI-II)
Description: Beck Depression Inventory II ranges from 0-63. Higher score indicates more severe depression. 0-13 minimal depression, 14-19 mild depression, 20-28 moderate depression, 29-63 severe depression.
Time Frame: from the beginning (0 weeks) to end (12 weeks) of the double-blind phase
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Change in BDI-II score
Arm/Group | Paroxetine | Venlafaxine Extended Release | Placebo
Number analyzed (Participants) | 42 | 34 | 39
Change in BDI-II score | -9.7 (1.1) | -9.6 (1.2) | -5.2 (1.1)

4. Secondary Outcome: Change in Geriatric Depression Rating Scale (GDS)
Description: Geriatric Depression Scale ranges from 0-30. Higher score indicates more severe depression. 0-9 normal, 10-19 mild depression, 20-30 severe depression.
Time Frame: from the beginning (0 weeks) to end (12 weeks) of the double-blind phase
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Change in GDS score
Arm/Group | Paroxetine | Venlafaxine Extended Release | Placebo
Number analyzed (Participants) | 42 | 34 | 39
Change in GDS score | -6.9 (1.0) | -6.9 (1.1) | -2.8 (1.0)

5. Secondary Outcome: Change in Brief Psychiatric Rating Scale (BPRS)
Description: Brief Psychiatric Rating Scale. Maximum score 126. Higher score indicates greater psychiatric difficulties.
Time Frame: from the beginning (0 weeks) to end (12 weeks) of the double-blind phase
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Change in BPRS score
Arm/Group | Paroxetine | Venlafaxine Extended Release | Placebo
Number analyzed (Participants) | 42 | 34 | 39
Change in BPRS score | -9.0 (1.3) | -9.8 (1.4) | -4.4 (1.3)

6. Secondary Outcome: Change in Unified Parkinson's Disease Rating Scale (UPDRS)
Description: Unified Parkinson's Disease Rating Scale. Higher score indicates more severe Parkinson's disease symptoms. Total maximum = 176. Mental maximum = 52, Activities of Daily Living maximum = 52, Motor maximum = 72. Minimum = 0.
Time Frame: from the beginning (0 weeks) to end (12 weeks) of the double-blind phase
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Change in UPDRS score
Arm/Group | Paroxetine | Venlafaxine Extended Release | Placebo
Number analyzed (Participants) | 42 | 34 | 39
Change in UPDRS score | -8.7 (2.1) | -7.0 (2.3) | -4.3 (2.0)

7. Secondary Outcome: Change in Snaith Clinical Anxiety Scale (CAS)
Description: Snaith Clinical Anxiety Scale. Range 0-21. Higher scores indicate increased anxiety. Score greater than 8 indicates clinical anxiety.
Time Frame: from the beginning (0 weeks) to end (12 weeks) of the double-blind phase
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Change in CAS score
Arm/Group | Paroxetine | Venlafaxine Extended Release | Placebo
Number analyzed (Participants) | 42 | 34 | 39
Change in CAS score | -3.6 (0.6) | -3.2 (0.6) | -2.4 (0.6)

8. Secondary Outcome: Change in Pittsburgh Sleep Quality Index (PSQI)
Description: Pittsburgh Sleep Quality Index scores range from 0-21, with higher scores indicating severe sleep difficulties.
Time Frame: from the beginning (0 weeks) to end (12 weeks) of the double-blind phase
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Change in PQSI score
Arm/Group | Paroxetine | Venlafaxine Extended Release | Placebo
Number analyzed (Participants) | 42 | 34 | 39
Change in PQSI score | -2.1 (0.4) | -2.6 (0.5) | -1.1 (0.4)

9. Secondary Outcome: Change in Unified Parkinson's Disease Rating Scale (UPDRS) - Motor
Description: Unified Parkinson's Disease Rating Scale - Motor has a maximum score of 72, minimum score of 0. Higher score indicates more severe Parkinson's disease symptoms.
Time Frame: from the beginning (0 weeks) to end (12 weeks) of the double-blind phase
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Change in UPDRS-motor score
Arm/Group | Paroxetine | Venlafaxine Extended Release | Placebo
Number analyzed (Participants) | 42 | 34 | 39
Change in UPDRS-motor score | -4.3 (1.5) | -2.0 (1.6) | -1.0 (1.5)

10. Secondary Outcome: Change in Unified Parkinson's Disease Rating Scale (UPDRS) - Tremor
Description: Unified Parkinson's Disease Rating Scale - Tremor subscale ranges from 0-23. Higher score indicates more severe Parkinson's disease symptoms.
Time Frame: from the beginning (0 weeks) to end (12 weeks) of the double-blind phase
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Change in UPDRS-tremor score
Arm/Group | Paroxetine | Venlafaxine Extended Release | Placebo
Number analyzed (Participants) | 42 | 34 | 39
Change in UPDRS-tremor score | 0.4 (0.5) | 0.5 (0.5) | -0.6 (0.5)

11. Secondary Outcome: Change in Unified Parkinson's Disease Rating Scale (UPDRS) - Bulbar
Description: Unified Parkinson's Disease Rating Scale - Bulbar maximum score 24, minimum score of 0. Higher score indicates more severe Parkinson's disease symptoms.
Time Frame: from the beginning (0 weeks) to end (12 weeks) of the double-blind phase
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Change in UPDRS-Bulbar score
Arm/Group | Paroxetine | Venlafaxine Extended Release | Placebo
Number analyzed (Participants) | 42 | 34 | 39
Change in UPDRS-Bulbar score | -1.4 (0.3) | -1.4 (0.3) | -0.5 (0.3)

12. Secondary Outcome: Change in Parkinson's Disease Questionnaire (PDQ) - 39 - Overall
Description: Parkinson's Disease Questionnaire (PDQ-39) Total. Range 0-100. Lower score indicates a better perceived health status.
Time Frame: from the beginning (0 weeks) to end (12 weeks) of the double-blind phase
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Change in PDQ-39 score
Arm/Group | Paroxetine | Venlafaxine Extended Release | Placebo
Number analyzed (Participants) | 42 | 34 | 39
Change in PDQ-39 score | -8.0 (2.3) | -8.4 (2.4) | -5.3 (2.1)

13. Secondary Outcome: Change in Parkinson's Disease Questionnaire (PDQ) - 39 - Emotional Well-Being
Description: Parkinson's Disease Questionnaire (PDQ-39) - Emotional Well-Being maximum score 24, minimum score of 0.Lower score indicates a better perceived health status.
Time Frame: from the beginning (0 weeks) to end (12 weeks) of the double-blind phase
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Change in PDQ-39 Emotional score
Arm/Group | Paroxetine | Venlafaxine Extended Release | Placebo
Number analyzed (Participants) | 42 | 34 | 39
Change in PDQ-39 Emotional score | -21.4 (3.3) | -20.7 (3.5) | -10.9 (3.1)

14. Secondary Outcome: Change in Short Form 36 Health Survey - Mental Component Summary
Description: Short Form 36 Health Survey. Range 0-100. Higher score indicates a better perceived quality of life.
Time Frame: from the beginning (0 weeks) to end (12 weeks) of the double-blind phase
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Change in SF-36 mental score
Arm/Group | Paroxetine | Venlafaxine Extended Release | Placebo
Number analyzed (Participants) | 42 | 34 | 39
Change in SF-36 mental score | 11.4 (1.7) | 9.5 (1.8) | 4.8 (1.6)

15. Secondary Outcome: Change in Short Form 36 Health Survey - Vitality
Description: Short Form 36 Health Survey - Vitality subscale ranges from 0-100. Higher score indicates a better perceived quality of life.
Time Frame: from the beginning (0 weeks) to end (12 weeks) of the double-blind phase
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Change in SF-36 vitality score
Arm/Group | Paroxetine | Venlafaxine Extended Release | Placebo
Number analyzed (Participants) | 42 | 34 | 39
Change in SF-36 vitality score | 13.5 (3.1) | 9.1 (3.3) | 4.7 (2.9)

16. Secondary Outcome: Change in Short Form 36 Health Survey - Role-Emotional
Description: Short Form 36 Health Survey - Emotional subscale ranges from 0-100. Higher score indicates a better perceived quality of life.
Time Frame: from the beginning (0 weeks) to end (12 weeks) of the double-blind phase
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Change in SF-36 Role score
Arm/Group | Paroxetine | Venlafaxine Extended Release | Placebo
Number analyzed (Participants) | 42 | 34 | 39
Change in SF-36 Role score | 39.5 (7.5) | 26.9 (8.0) | 12.7 (6.9)

17. Secondary Outcome: Change in Short Form 36 Health Survey - Mental Health
Description: Short Form 36 Health Survey - Mental Health subscale ranges from 0-100. Higher score indicates a better perceived quality of life.
Time Frame: from the beginning (0 weeks) to end (12 weeks) of the double-blind phase
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Change in SF-36 Mental Health score
Arm/Group | Paroxetine | Venlafaxine Extended Release | Placebo
Number analyzed (Participants) | 42 | 34 | 39
Change in SF-36 Mental Health score | 16.7 (2.7) | 17.4 (2.8) | 9.7 (2.5)

ADVERSE EVENTS:
Arm/Group | Paroxetine | Venlafaxine Extended Release | Placebo
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/34 | 0/39
Other Adverse Events (participants affected / at risk) | 10/42 | 8/34 | 9/39
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paroxetine (N=42) | Venlafaxine Extended Release (N=34) | Placebo (N=39)
Insomnia (Psychiatric disorders) | 1 (1) | 7 (7) | 9 (9)
Abnormal Dreaming (Psychiatric disorders) | 1 (1) | 1 (1) | 4 (4)
Somnolence (Psychiatric disorders) | 8 (8) | 8 (8) | 5 (5)
Diaphoresis (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (4) | 4 (4)
Pruritis (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 6 (6) | 7 (7) | 5 (5)
Nausea (Gastrointestinal disorders) | 6 (6) | 5 (5) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 3 (3) | 3 (3)
Sexual Dysfunction (Reproductive system and breast disorders) | 10 (10) | 8 (8) | 4 (4)
Fatigue (General disorders) | 9 (9) | 4 (4) | 5 (5)
Back Pain (General disorders) | 0 (0) | 2 (2) | 1 (1)
Chest Pain (General disorders) | 0 (0) | 2 (2) | 0 (0)
Hot Flushes (General disorders) | 0 (0) | 0 (0) | 2 (2)
Tremor (Nervous system disorders) | 7 (7) | 7 (7) | 3 (3)
Dyskinesia (Nervous system disorders) | 1 (1) | 4 (4) | 3 (3)
Dizziness (Nervous system disorders) | 7 (7) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 6 (6) | 8 (8) | 6 (6)
Balance Difficulty (Nervous system disorders) | 2 (2) | 3 (3) | 3 (3)
Numbness/Parasthesia (Nervous system disorders) | 3 (3) | 1 (1) | 4 (4)
Parkinsonism Aggravated (Nervous system disorders) | 3 (3) | 5 (5) | 4 (4)
Hypertension (Cardiac disorders) | 1 (1) | 4 (4) | 0 (0)
Micturition Difficulty (Renal and urinary disorders) | 5 (5) | 1 (1) | 1 (1)
Weight Gain (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (2)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2)
Agitation (Psychiatric disorders) | 0 (0) | 2 (2) | 3 (3)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 5 (5)
Irritability (Psychiatric disorders) | 1 (1) | 2 (2) | 6 (6)
Decreased Libido (Psychiatric disorders) | 3 (3) | 5 (5) | 2 (2)
Marked Restlessness (Psychiatric disorders) | 3 (3) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No